CLINICAL TRIAL: NCT05961410
Title: Eltrombopag Plus G-CSF for Human CD34+ Cell Mobilization in Patients With Lymphoma Undergoing Autologous Stem Cell Harvest
Brief Title: Eltrombopag for Peripheral Blood Stem Cell Harvest
Acronym: EPBSCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202301091MIFC
Record Dates: First submitted 2023-07-09; First posted 2023-07-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma; Peripheral Blood Stem Cell Transplantation
Keywords: Lymphoma; Peripheral Blood Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eltrombopag (Experimental): ESHAP + Eltrombopag as peripheral blood stem cell mobilization
  Interventions: Drug: Eltrombopag olamine

INTERVENTIONS:
Drug: Eltrombopag olamine — Patients will receive eltrombopag 75 mg/day from ESHAP D6 until end of stem cell harvest.
  Other Names: Revolade

SUMMARY:
The goal of this clinical trial is to explore the activity of eltrombopag in lymphoma patients receiving autologous hematopoietic stem cell harvest. The main questions it aims to answer are:

* Determine the efficacy of adding eltrombopag during autologous hematopoietic stem cell mobilization and harvest.
* Determine the pharmacokinetics and pharmacodynamics of serum eltrombopag concentration, circulating CD34+ cells during autologous hematopoietic stem cell mobilization.

Participants will receiving additional eltrombopag during stem cell harvest procedure. The amount of harvested stem cells will be compared with historical group to see if eltrombopag could increase the amount of harvested stem cells.

DETAILED DESCRIPTION:
Autologous hematopoietic stem cell transplantation (auto-HSCT) is the standard treatment for many malignant diseases, including plasma cell myeloma, lymphoma and germ-cell tumor. In the USA, it is estimated that 34,920 new cases of myeloma, 81,560 new cases of non-Hodgkin lymphoma, and 8830 new cases of Hodgkin lymphoma will be diagnosed annually.

Auto-HSCT is the first line therapy for fit patients with plasma cell myeloma and second line therapy for fit patients with relapsed/refractory lymphoma. It significantly prolongs overall survival in patients with myeloma and provides chances of cure in patients with relapsed/refractory lymphoma. The prerequisite condition to successfully perform an auto-HSCT is to mobilize and harvest an adequate amount of autologous hematopoietic stem cells. Usually, a number of 0.75-2.5 x 10^6/kg CD34+ cell is the minimal amount of hematopoietic stem cells required to safely perform an auto-HSCT. Recent study revealed increased amount of CD34+ autologous hematopoietic stem cell dose in auto-HSCT as a predictor of shortened engraftment time and better survival.

Before PBSC (peripheral blood stem cell) harvest, the hematopoietic stem cells need to be mobilized from bone marrow into the peripheral blood. In patients with malignant diseases, chemo-mobilization is the preferred mobilization method, which consists of chemotherapy 1-2 weeks prior to the harvesting procedure. Granulocyte colony-stimulating factor (G-CSF) is administered after the chemotherapy to facilitate PBSC mobilization. Following chemotherapy and G-CSF, PBSC will be mobilized into peripheral blood for harvest. The concentration of PBSC will be monitored. Once an adequate amount of PBSC is measured, a PBSC harvest procedure will be initiated. The PBSC harvest procedure usually starts 1-2 weeks following chemotherapy, and takes 1-5 days until adequate amounts of PBSC are collected. The more days a harvesting procedure takes, the larger medical risks and costs it possesses.

ESHAP is one of the most commonly used chemo-mobilization regimens in National Taiwan University Hospital. The unpublished data from National Taiwan University Hospital revealed that, it took at least 2 days to obtain adequate amount of PBSC for auto-HSCT in 40.84% of patients.

Under certain circumstances, patients may never obtain adequate amounts of PBSC for auto-HSCT even after 5 days of PBSC harvest or salvage treatment with plerixafor, a stem cell mobilizer agent. Compared to patients who obtained an adequate amount PBSC in the 1st day of stem cell harvest, these patients undertook more risks during harvest procedure and cost more medical expenditure. In addition, plerixafor is an expensive medication ($9,255 USD/each supply) that is conditional reimbursed in Taiwan. It is likely to be unaffordable for patients outside Taiwan or those without reimbursement. Without adequate amounts of harvested stem cells, the standard treatment of lymphoma (auto-HSCT) can't be performed and patient's outcome will be severely compromised. There's an urgent need to increase the percentage of patients gathering an adequate amount of PBSC on the first harvest day.

Eltrombopag is a thrombopoietin (TPO) receptor agonist that has been approved by the United States Food and Drug Administration for the treatment of immune thrombocytopenia (2007) and aplastic anemia (2014). It has been proven that TPO agonists can stimulate stem cell proliferation and maintenance. One study showed administration of eltrombopag increased the stem cell amount harvested from patients with plasma cell myeloma. Investigators hypothesized that addition of eltrombopag during ESHAP PBSC mobilization will increase the amount of harvested stem cells in patients with lymphoma.

In addition, a study in patients with aplastic anemia showed positive correlation of serum eltrombopag concentration with treatment efficacy. A higher peak serum eltrombopag concentration were associated with higher response rate. This raises the interest of measuring serum eltrombopag in this study. The association of serum eltrombopag concentration and harvested PBSC amount will be explored as well.

In conclusion, this study aimed to explore the activity of eltrombopag in ESHAP PBSC mobilization. Participants will receive eltrombopag following ESHAP chemo-mobilization. The amount of PBSC, and its association with peak serum eltrombopag will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Diagnosis: Hodgkin lymphoma or non-Hodgkin lymphoma
* Disease status: complete response, partial response, or stable disease after at least 2 cycles of treatment (see appendix 2 for definition)
* Planned to receive ESHAP (etoposide, steroid, high-dose cytarabine, cisplatin) chemotherapy with/without monoclonal antibody (ex: rituximab, brentuximab) as chemo-mobilization for stem cell harvest
* East-Asian heritage

Exclusion Criteria:

* History of vascular thromboembolic event
* Steady state platelet count > 1000k/μL
* Documented cytogenetic abnormalities in marrow blood
* Current administration of eltrombopag
* History of grade III-IV hepatotoxicity to eltrombopag 75/mg/day
* Life-threatening allergic reactions to eltrombopag
* Baseline serum aspartate aminotransferase (AST), alanine aminotransferase(ALT) or total bilirubin > 3 fold of upper limit of normal
* Pregnancy or breast-feeding
* Patients with hepatitis C receiving interferon and ribavirin treatment
* Concurrent active cancer other than lymphoma
* Eastern Cooperative Oncology Group (ECOG) 3-4 (see appendix 4 for definition)
* Moribund status such as concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious disease that death within 30 days is likely.
* Inability to understand the investigational nature of the study or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of harvested CD34+ cells in first stem cell harvest day | 1 day (first stem cell harvest day)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 8 months
Engraftment time (days) of granulocytes | Whole hematopoietic stem cell transplantation process, an average of 4 weeks
  The time needed to achieve absolute neutrophil count > 500 x 10^6/L after stem cell infusion in study participants
Engraftment time (days) of platelets | Whole hematopoietic stem cell transplantation process, an average of 4 weeks
  The time needed to achieve platelet > 20,000/L without transfusion after stem cell infusion in study participants
Peak serum eltrombopag concentration | 3 weeks
  Peak serum eltrombopag concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Chuan Yu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shpall EJ, Champlin R, Glaspy JA. Effect of CD34+ peripheral blood progenitor cell dose on hematopoietic recovery. Biol Blood Marrow Transplant. 1998;4(2):84-92. doi: 10.1053/bbmt.1998.v4.pm9763111.
- [Background] Zuo W, Zhang B, Ruan J, Chen M, Han B. Correlation of the Plasma Concentration of Eltrombopag With Efficacy in the Treatment of Refractory Aplastic Anemia: A Single-Centre Study in China. Front Pharmacol. 2020 Nov 16;11:582625. doi: 10.3389/fphar.2020.582625. eCollection 2020. PMID 33364958
- [Background] Zhu J, Hao SG, Hu J, Zhuang JL, Wang C, Bai HT. rhTPO combined with chemotherapy and G-CSF for autologous peripheral blood stem cells in patients with refractory/relapsed non-Hodgkin's lymphoma. Cancer Manag Res. 2019 Sep 13;11:8371-8377. doi: 10.2147/CMAR.S219242. eCollection 2019. PMID 31571993
- [Background] Scheinberg P. Activity of eltrombopag in severe aplastic anemia. Blood Adv. 2018 Nov 13;2(21):3054-3062. doi: 10.1182/bloodadvances.2018020248. PMID 30425070